CLINICAL TRIAL: NCT06786013
Title: Effects of Interscalene Block Anesthesia on Visual Clarity and Hemodynamic Parameters in Arthroscopic Rotator Cuff Repair: A Prospective, Randomized Study
Brief Title: Effects of Interscalene Block on Visual Clarity in Arthroscopic Surgery
Status: Completed | Type: Observational
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Alper Kilicaslan, Alper Kılıçaslan, MD, Prpf, Specialist in Anesthesiology and Reanimation., Konya Necmettin Erbakan Üniversitesi
Other Study IDs: 2024/5217
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Syndrome
Keywords: interscalene block; visual clarity; Arthroscopic rotator cuff repair

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interscalene brachial plexus block (ISB): The group that received ISB for arthroscopic rotator cuff repair anesthesia
- General anesthesia group: The group that received general anesthesia for arthroscopic rotator cuff repair

SUMMARY:
Arthroscopic rotator cuff repair (RCR) has become the predominant technique for managing patients with full-thickness rotator cuff tears. Optimizing visual clarity is crucial for performing shoulder arthroscopy safely, precisely, and successfully. However, intraoperative bleeding remains the most significant factor impairing visual clarity.

The interscalene brachial plexus block (ISB) technique is widely employed in shoulder joint and upper extremity surgeries. However, ISB may lead to hypertension due to the spread of local anesthetic to adjacent structures, such as the carotid sinus baroreceptors. Hypertension-induced microbleeding can obstruct the surgical field of view.

Our hypothesis suggests that arthroscopic visual clarity may be compromised in awake patients receiving ISB for anesthesia.

This study aims to compare the effects of interscalene brachial plexus block and general anesthesia on hemodynamic parameters and visual clarity in patients undergoing arthroscopic rotator cuff repair surgery.

DETAILED DESCRIPTION:
Our study will be conducted prospectively, and no additional medication or interventional procedure will be administered to the patients. A total of 80 patients, 40 from the general anesthesia group and 40 from the interscalene block anesthesia group, who meet the inclusion criteria, will be included in the study. In both groups, systolic arterial blood pressure (SAB), diastolic arterial blood pressure (DAB), mean arterial blood pressure (MAP), and heart rate (HR) values will be recorded every 5 minutes throughout the operation after the surgical procedure begins. At the end of the operation, visual clarity will be assessed by the same surgeon (M.O) using a Numeric Rating Scale (0 = very poor, 10 = excellent). To detect a 2-point (20%) difference in the NRS score for visual clarity, a total of 37 patients are required with 80% power and a significance level of 0.05. This calculation assumes that such an effect is clinically significant and that the standard deviation is 2.21. Assuming a 10% dropout rate, we calculated that a total of 80 patients would be needed for two groups, with 40 patients per group.

Descriptive statistics, including mean, standard deviation, median, minimum, maximum, frequency, and percentage, will be used to summarize the data. The Kolmogorov-Smirnov test will be employed to assess the distribution of variables. For the comparison of quantitative data, the Independent Samples t-test and Mann-Whitney U test will be utilized. For the comparison of qualitative data, the Chi-Square test will be used. A p-value less than 0.05 will be considered statistically significant.

The cut-off values of quantitative parameters will be determined using ROC analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to provide informed consent.
* Patients able to reliably report their symptoms to the research team.
* ASA physical status classification of 1-3.
* Scheduled to undergo arthroscopic rotator cuff repair surgery in the lateral decubitus position.

Exclusion Criteria:

* Contraindications to anesthesia.
* Patients under 18 years old.
* Cognitive impairment or communication barriers.
* BMI > 40.
* Weight less than 50 kg or more than 100 kg.
* Psychiatric disorders.
* Chronic opioid therapy for pain.
* Severe liver, heart, or kidney failure.
* Hypertension (possibly severe, depending on the study context).
* Use of opioids for any reason.
* Revision shoulder surgery.
* Diaphragmatic paralysis on the opposite side of the planned intervention.
* Concurrent anticoagulation therapy or coagulopathy.
* Skin deformities or infections in the block area.
* Progressive neurological deficits affecting peripheral nerves.
* Allergy to amide-structured local anesthetics.
* ASA physical classification score ≥4.
* Suspected or confirmed pregnancy.
* Breastfeeding mothers.
* Patients who do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo arthroscopic rotator cuff repair
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Visual clarity during arthroscopic rotator cuff repair | 1 day
  Visual clarity of the arthroscopic view will be assessed by the same surgeon (MO) using a Numeric Rating Scale (0 = very poor, 10 = excellent).

SECONDARY OUTCOMES:
Hemodynamic parameters | 1 day
  systolic arterial blood pressure (mm Hg), diastolic arterial blood pressure (mm Hg), mean arterial blood pressure (mm Hg), and heart rate (beats per minute) values will be recorded every 5 minutes after IS block and throughout the surgery pressure (mm/Hg), and heart rate (beats per minute) values will be recorded every 5 minutes throughout the operation
Visual analog scale (VAS) pain scores | at 6,12, 18, 24 hours postoperatively
  Pain was evaluated by blinded researcher using visual analog scale (VAS) pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Alper KILICASLAN, Prof, Principal Investigator — Konya Necmettin Erbakan Universty Medical Faculty /Türkiye
Locations (1):
- Alper Kilicaslan, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gianesello L, Magherini M, Pavoni V, Horton A, Nella A, Campolo MC. The influence of interscalene block technique on adverse hemodynamic events. J Anesth. 2014 Jun;28(3):407-12. doi: 10.1007/s00540-013-1748-8. Epub 2013 Nov 21. PMID 24258467
- [Result] Bildik C, Pehlivanoglu T. Arthroscopic rotator cuff repair performed with intra-articular tranexamic acid: could it provide improved visual clarity and less postoperative pain? A prospective, double-blind, randomized study of 63 patients. J Shoulder Elbow Surg. 2023 Feb;32(2):223-231. doi: 10.1016/j.jse.2022.10.007. Epub 2022 Nov 18. PMID 36403924